CLINICAL TRIAL: NCT06469697
Title: Utilizing Traditional and Modern Music Performance in Eye Health Education to Improve Child Eye Health Service Uptake in Zanzibar
Brief Title: Zanzibar Arts for Children's Eyesight Pilot Trial
Acronym: ZANZI-ACEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Ministry of Health and Social Welfare, Zanzibar (Other Government)
Responsible Party: Principal Investigator, Ving Fai Chan, Senior Lecturer, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHLS 23_32
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Myopia; Conjunctivitis; Hyperopia
Keywords: Arts; Health education; Refractive errors; Conjunctivitis
MeSH Terms: conditions — Myopia; Conjunctivitis; Hyperopia; Arts syndrome; Health Education; Refractive Errors

STUDY DESIGN:
Intervention Model Description: This is pilot will be conducted in 9 schools where radio broadcasts and community broadcasts will be implemented (intervention) and 9 schools where only community broadcasts will be implemented (comparator).
Who Masked: Care Provider
Masking Description: Care providers will not be able to know whether the children referred are from intervention not comparator group as they will only receive a generic referral form from the project.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Musical pieces developed by the Ministry of Education and Vocational Training will be played at intervention schools using compact discs. These will be broadcast once during morning assembly, once during recess, and once before school ends on Mondays and Fridays for 3 months. After this period, a popular local radio station will broadcast the music pieces three times a day during peak hours.
  Interventions: Behavioral: School music broadcast
- Comparator (Active Comparator): A popular local radio station will broadcast the music pieces three times a day during peak hours, coinciding with the times when the intervention group is receiving the same program (community broadcast).
  Interventions: Behavioral: Community music broadcast

INTERVENTIONS:
Behavioral: School music broadcast — An arts-based eye health intervention featuring traditional and contemporary music pieces will be broadcasted at both school and community levels.
  Arms: Intervention
Behavioral: Community music broadcast — An arts-based eye health intervention featuring traditional and contemporary music pieces will be broadcasted at community levels.
  Arms: Comparator

SUMMARY:
In Zanzibar, around 22,000 children (4% of those aged 6 to 12) need treatment for eye issues like conjunctivitis or require glasses. A 2017 study found that 42% of rural children needing glasses didn't have them. Many locals distrust Western medicine and prefer traditional remedies, rejecting public health efforts such as posters and brochures.

Globally, eye health promotion has been underfunded and overlooked. Research suggests community-designed interventions and behavior change studies are needed to promote sustainable eye health practices. Arts-based interventions using traditional storytelling and performances have been effective in Africa, improving health outcomes in areas like food hygiene and mental health. Health campaigns in schools might be less effective since parents make health decisions for their children.

This study aims to see how well using both traditional and modern music performances in an eye health education program can break down cultural barriers and increase children's use of eye health services in schools and communities. The investigators want to answer three main questions:

1. How effective is a 6-month music-based eye health education program in schools and communities at improving eye health knowledge and service use among parents and children?
2. What factors influenced the success of the 6-month music-based eye health education program?
3. What are the costs and benefits of this 6-month program in increasing eye health service use among children in schools and communities?

DETAILED DESCRIPTION:
Problem: Zanzibar has about 22,000 children (4% of 6-to-12-year-old children) needing conjunctivitis treatment or spectacle correction (Ministry of Health, unpublished report). A 2017-case study showed that about 42% of children in rural Zanzibar communities who needed a pair of glasses did not have them.(1) Local stakeholders engagement revealed that underlying suspicions of Western medicine and public health initiatives led people to continue using traditional, less effective healing methods. Although health posters and brochures have successfully increased service uptake in other contexts,(2) our engagement with stakeholders revealed rejection of such initiatives among the Zanzibari community, such as when the posters were removed or vandalized.

Worldwide, eye health promotion has received limited attention and funding.(2) A Cochrane review(3) and The Lancet Global Health Commission on Global Eye Health(4) suggested that behavior change and co-design studies are needed to provide evidence on promoting sustainable behavior changes among the community and children with eye problems. Health-focused arts-based interventions have been shown to catalyze behavioral changes in Africa because they are built on traditional oral and performance methods.(5) A review(6) has shown that traditional music incorporated into health promotion campaigns to improve food hygiene, perinatal mental health and Ebola in Gambia yielded highly positive results. Less effective may be health promotion strategies implemented in school settings only because parents are the ultimate decision-makers of health choices for their children.

Research questions: The study aims to explore "the effectiveness of utilizing traditional and modern music performances in an eye health education strategy implemented in school and community settings to reduce socio-cultural barriers and subsequently increase child eye health service uptake". The specific research questions are:

1. How effective is a 6-month arts-based eye health education strategy implemented in school and community settings to improve parents' and children's eye health literacy and eye service uptake?
2. Which factors influenced the uptake of the 6-month arts-based eye health education strategy?
3. What are the cost and benefits of a 6-month arts-based eye health education strategy on improving eye health service uptake among children in school and community settings?

A: Assess the effectiveness of a 6-month arts-based eye health education program implemented in school and then community settings to improve parents' and children's eye health literacy and eye service uptake

1. Trained teachers will screen approximately 8000 children in eight intervention schools (with art-based eye health education program) and eight control schools (without any health education program) and refer approximately 400 children with vision <6/12 or/and refractive error (RE) and obvious eye diseases for free ocular management at the local eye clinics (current practice). Teachers in enrolled schools will maintain an eye health register to record the names of children who failed vision screening tests and are then referred for treatment, the reasons for referral, and follow up on which children attended an eye examination at the referral clinics. With an estimated prevalence of children with refractive error and obvious eye diseases of 5%, the investigators will have a sufficient sample size for analysis in this pilot trial.
2. Before the intervention, the investigators will administer a baseline demographic profile survey to all 400 children with refractive error and obvious eye diseases and their parents, 400 children with normal vision and their parents, followed by a baseline knowledge and attitude survey. Children referred for further ocular management will be followed up at Month 3 to determine the proportion of them who have gone for an eye examination at the hospital (baseline uptake rate). The enrolment will begin in Month 4. Subsequently, the eye health education will be broadcasted at intervention schools once during morning assembly, once during recess and once before school on Monday and Friday starting at Month 4. At Month 10, the endline 1 data (children's knowledge and attitude survey, eye health register checks) will be collected to determine follow-up scores and rates.
3. At Month 11, a popular local radio station will broadcast eye health education in the musical form three times a day. At Month 14, the second follow-up data (parents' knowledge and attitude survey, eye health register checks) will be collected to determine endline 2 follow-up scores/rates.
4. The primary outcomes are the change in the proportion of children accessing eye health services and the change in children's and parents' knowledge and attitude scores from baseline and endline 1 and endline 2. The secondary outcomes are the proportion and causes of children failing eye health screening, the proportion of children wearing spectacles during an unannounced visit and the children's self-reported compliance to eye medication treatment.

B: Explore in what ways social, cultural and artistic factors influenced the uptake of the arts-based eye health education strategy

1. Stakeholders involved in the music pieces' co-creation process will be invited to identify and reflect on the achievements, gaps, and barriers between what was intended by them and what was received by the intended audience. Stakeholders include Ministries' representatives, community and religious leaders, artist groups, parents, children, teachers and traditional healers. Semi-structured interviews will be conducted 6 months after the program implementation.
2. A series of small group discussions and individual interviews will be held with various target audiences of the intervention to ascertain responses to the intervention by those not involved in its design. These will include children, their guardians, teachers, health care practitioners, traditional healers, radio broadcasters and cultural workers from the context to determine 'audience reception'.
3. Thematic analysis will be conducted to ascertain (i) the efficacy of the makers' intentionality for the intervention concerning the reception of the pieces in context ('fitness-for-purpose'); (ii) the conceptual impact of the content of the music pieces in terms of the socio-cultural barriers addressed and myths dispelled, and how this intervention has contributed to new and/or existing counter-narratives of eye health; (iii) the reception of the music form of the pieces, including associated with past (heritage), current and aspirational (contemporary) genres and registers, and in what ways such artistic and cultural associations have contributed to the intervention's efficacy.

C: Determine the cost and benefits of a short-term arts-based eye health education strategy on improving eye health service uptake among children to inform upscale investment decisions

1. The investigators will develop a costing tool to (i) identify the main implementing costs, including the time and skills to develop the radio broadcast; (ii) calculate the costs of the intervention's roll-out to schools and the wider community; (iii) determine the costs that the intervention may save in the longer term, such as from absenteeism or treatment made unnecessary because of early treatment.
2. The pilot will enable us to cost the intervention and how affordable it is. By looking at the uptake of the intervention in schools and the community, the investigators can compare the costs and benefits of the strategies. Value is defined as cost relative to benefits, whereas budget impact is about costs only. Both are widely used for healthcare investment decisions in LMIC. This will enable policymakers to assess how affordable the intervention is. Understanding what are given up when a new intervention is funded (what else could have done with these resources) and the return on investment is crucial to helping policymakers decide whether the program is worth the investment.

ELIGIBILITY:
Inclusion Criteria:

* primary and secondary schools with student school-going rates of approximately 75%
* schools with similar number of boys and girls
* schools within 5km of the nearest eye centres.
* school children who have either an obvious eye disease tested using a pen torch test and/or a presenting distance visual acuity ≤6/12 in either eye, and their parents.

Exclusion Criteria:

* primary and secondary schools with student school-going rates of less than 75%
* schools with imbalance number of boys and girls
* schools above 5km of the nearest eye centres.
* school children who do not have either an obvious eye disease tested using a pen torch test and/or a presenting distance visual acuity ≤6/12 in either eye, and their parents.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1295 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of children accessing eye health services | Three months and six months after the intervention is implemented
  Proportion of children who have gone for eye treatment at the referral sites over those who failed eye health screening and referred to the referral site; measured in percentage, the higher the percentage the better the referral rate

SECONDARY OUTCOMES:
Children spectacle compliance | Three months and six months after the intervention is implemented
  Possession of glasses at school during an unannounced examination will be measured as either yes or no. A higher proportion of "yes" responses indicates better compliance.
Children eye drops usage compliance | Three months and six months after the intervention is implemented
  Self-reported completion of eye drop treatment will be measured as either yes or no. A higher proportion of "yes" responses indicates better compliance.
Cost-benefit analysis | Through study completion, 6 months after the intervention is implemented.
  Costs will be measured by the program expenses, while benefits will be assessed by the proportion of children who voluntarily seek eye treatment at referral sites compared to those who failed the eye health screening and were referred. A higher proportion of treated children per US dollar spent indicates a higher cost-benefit ratio.
Parents knowledge and attitude | Three months and six months after the intervention is implemented
  A 27-item questionnaire will be used for measurement. Each question requires a yes or no response. A higher number of "yes" answers indicates better knowledge and attitude.
Children's knowledge and attitude | Three months and six months after the intervention is implemented
  A 27-item questionnaire will be used for measurement. Each question requires a yes or no response. A higher number of "yes" answers indicates better knowledge and attitude.
Cost effectiveness analysis | Through study completion, 6 months after the intervention is implemented.
  Cost will be measured by the program expenses, while effectiveness will be assessed using the Visual Analogue Scale (EQ-5Q-Y questionnaire). A higher score per US dollar indicates greater cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Ving Fai Chan, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Ministry of Health, Zanzibar, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hobday K, Ramke J, du Toit R. Eye health promotion in Western Pacific island countries. Clin Exp Ophthalmol. 2011 Aug;39(6):584-5. doi: 10.1111/j.1442-9071.2011.02514.x. No abstract available. PMID 21631663
- [Background] Evans JR, Morjaria P, Powell C. Vision screening for correctable visual acuity deficits in school-age children and adolescents. Cochrane Database Syst Rev. 2018 Feb 15;2(2):CD005023. doi: 10.1002/14651858.CD005023.pub3. PMID 29446439
- [Background] Burton MJ, Ramke J, Marques AP, Bourne RRA, Congdon N, Jones I, Ah Tong BAM, Arunga S, Bachani D, Bascaran C, Bastawrous A, Blanchet K, Braithwaite T, Buchan JC, Cairns J, Cama A, Chagunda M, Chuluunkhuu C, Cooper A, Crofts-Lawrence J, Dean WH, Denniston AK, Ehrlich JR, Emerson PM, Evans JR, Frick KD, Friedman DS, Furtado JM, Gichangi MM, Gichuhi S, Gilbert SS, Gurung R, Habtamu E, Holland P, Jonas JB, Keane PA, Keay L, Khanna RC, Khaw PT, Kuper H, Kyari F, Lansingh VC, Mactaggart I, Mafwiri MM, Mathenge W, McCormick I, Morjaria P, Mowatt L, Muirhead D, Murthy GVS, Mwangi N, Patel DB, Peto T, Qureshi BM, Salomao SR, Sarah V, Shilio BR, Solomon AW, Swenor BK, Taylor HR, Wang N, Webson A, West SK, Wong TY, Wormald R, Yasmin S, Yusufu M, Silva JC, Resnikoff S, Ravilla T, Gilbert CE, Foster A, Faal HB. The Lancet Global Health Commission on Global Eye Health: vision beyond 2020. Lancet Glob Health. 2021 Apr;9(4):e489-e551. doi: 10.1016/S2214-109X(20)30488-5. Epub 2021 Feb 16. No abstract available. PMID 33607016
- [Background] McConnell BB. Music and health communication in The Gambia: A social capital approach. Soc Sci Med. 2016 Nov;169:132-140. doi: 10.1016/j.socscimed.2016.09.028. Epub 2016 Sep 19. PMID 27721137
- [Derived] Omar F, Othman OJ, Yong AC, Belluigi D, Graham C, Graham R, Mashayo E, Chan VF. Preliminary effectiveness of musical messaging to improve child eye health service uptake in Zanzibar: a pilot randomised trial. BMJ Open. 2025 Sep 23;15(9):e107348. doi: 10.1136/bmjopen-2025-107348. PMID 40987737